CLINICAL TRIAL: NCT05733780
Title: A Phase 1b/2a Randomized, Blinded, Placebo-controlled Study in Participants With Mild to Moderate COVID-19 to Evaluate the Safety, Efficacy, and Pharmacokinetics of Orally Administered ProLectin-M
Brief Title: To Evaluate the Safety, Efficacy,and Pharmacokinetics of Orally Administered Prolectin-M
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bioxytran Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CTSRS/2205
Record Dates: First submitted 2022-12-26; First posted 2023-02-17 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: COVID-19; SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19 | interventions — galactomannan

STUDY DESIGN:
Intervention Model Description: A Phase 1b/2a Randomized, Blinded, placebo-controlled Study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding will be maintained throughout the trial until database is locked after last patient last visit. Emergency unblinding will be allowed through a 24/7 helpline set up for any investigator / ethics committee member or others authorized to request for unblinding. Given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): ProLectin M 1,400 mg Tab. Number of Doses -04 Dosing Frequency-once every 2 hours Total Dose/Day-5600 mg
  Interventions: Drug: Prolectin-M
- Arm 2 (Experimental): ProLectin M 1,400 mg Tab. Number of Doses -08 Dosing Frequency-Hourly Total Dose/Day-11200mg
  Interventions: Drug: Prolectin-M
- Arm 3 (Experimental): ProLectin M 1,400 mg Tab. Number of Doses -12 Dosing Frequency-Hourly Total Dose/Day-16800
  Interventions: Drug: Prolectin-M
- Arm 4 (No Intervention): Matching Placebo. Number of Doses -08 Dosing Frequency-Hourly Total Dose/Day-0 mg

INTERVENTIONS:
Drug: Prolectin-M — Prolectin-M
  Precise chemistry based molecule that binds to galectin like receptors on the N terminal of S1 subunit of the Sars-CoV2 virus
  Other Names: Galactomannan
  Arms: Arm 1; Arm 2; Arm 3

SUMMARY:
ProLectin M is an orally administered polysaccharide. Polysaccharides competitively bind to the N-terminal tail of human galectin-3 through a proline isomerization [10]. Galetin-3 (Gal-3) is 1 among the 15 galectins described in humans and also a ubiquitous human galectin expressed in various disease pathogenesis pathways [11].

The objective of this clinical study is to evaluate the safety and efficacy of a galectin antagonist, ProLectin M (a Guar Gum Galactomannan), in the treatment of subjects with asymptomatic to moderately-severe, ambulatory COVID-19 patients.

DETAILED DESCRIPTION:
This trial will test the efficacy of ProLectin M in lowering viral load among those infected with SARS-CoV-2. Viral load will be measured using nucleic acid amplification-based diagnostics, RT-PCR. The RT-PCR will measure an absolute increase in cycle threshold values from baseline.

ProLectin M (a guar gum galactomannan), an oral form of galectin antagonist could treat COVID-19 patients. When given early in the disease pathogenesis and the viral replication is stopped, it can prevent further spread of SARS-CoV-2 among the household contacts and their community.

ELIGIBILITY:
Inclusion Criteria:Patients must meet all of the following criteria to be included in this study.

1. Male or Female subject of ≥ 18 years of age, willing and able to provide written informed consent for participation in the study and ready to comply with the study procedures and schedule.
2. Subject having a positive diagnosis for presence of SARS-CoV- 2, obtained from a recently performed RT-PCR (≤ 3 days) with a Ct value ≤ 25.
3. Subject has the ability to take oral medication and be willing to adhere to the trial protocol regimen of repeated nasopharyngeal swab collections and follow up till day 14.
4. Females of child bearing potential who has been using a highly effective contraception for at least 1 month prior to screening and agrees to continue using it during the study participation/enrolment, confirmed through negative pregnancy test.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from this study.

1. Oxygen Saturation levels (SpO2) ≤ 94% on room air.
2. Female subjects who are pregnant or breastfeeding.
3. Subjects with any active malignancy or undergoing active chemotherapy.
4. Subjects who are currently receiving or have received any investigational treatment for COVID-19 within 30 days prior to screening.
5. Subjects with a history of hypercalcemia or serum calcium concentration >10mg/dl
6. Subjects currently on concomitant medication that can contains calcium, elevate serum calcium levels, or exacerbate hypercalcemia (Ex. Lithium, thiazide diuretics etc.).
7. Subjects currently on calcium-binding (chelation) concomitant medication that may result in reduction in absorption (e.g. fluroquinolone, bisphosphonates, antivirals such as integrase strand transfer inhibitors, antibiotics such as quinolones, tetracyclines etc.)
8. In the opinion of the Investigator, the participation of the subject in the study is not in the subject's best interest, or the subject has any medical condition that does not allow the study protocol to be followed safely.
9. Subjects with known allergies to any of the components used in the formulation of the interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Change In Clinical Status | Day 7
  Non-detection of viral shedding in nasopharyngeal swab detecting qualitative SARS-CoV-2

SECONDARY OUTCOMES:
Safety Outcome | from time of signing informed consent till day 14
  Proportion of participants with treatment-emergent AEs (TEAEs) and laboratory abnormalities.
Safety Outcome | from time of signing informed consent till day 14
  Proportion of participants with TEAEs leading to study treatment discontinuation
Mortality | from time of signing informed consent till day 14
  Mortality rate by Day 14
Plasma Concentration of PL-M | Day 7
  Characterization of the plasma concentrations of ProLectin-M and its metabolites including AUC0 24h, AUClast, CLss/F, t1/2, Vz/F, Cmax, Tmax, Clast, Tlast, AUCtau, λz, and Ctau
Time to discharge of viral load | from time of signing informed consent till day 14
  Time to negative SARS-CoV-2 polymerase chain reaction (PCR)
Change in Clinical Status from Baseline to End of the study | from time of signing informed consent till day 14
  Time to alleviation (absent) of baseline COVID- 19 symptoms as reported on the WHO clinical progression scale
Safety Outcome | from time of signing informed consent till day 14
  Rate of adverse events
Change in Clinical Status | Day 3 and Day 5
  Non-detection of viral shedding in nasopharyngeal swab detecting qualitative SARS-CoV-2 Outcome TimePoints Non-detection of viral shedding in nasopharyngeal swab detecting qualitative SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Sunitha Mali, Study Chair — Team Lead

IPD SHARING:
Plan to Share IPD: No
The sponsors and the study representatives and other stakeholders will take a decision on completion of the trial